CLINICAL TRIAL: NCT00673127
Title: A Phase II Trial of Ketoconazole, Hydrocortisone and Dutasteride in Asymptomatic Hormone Refractory Prostate Cancer
Brief Title: Ketoconazole, Hydrocortisone and Dutasteride in Asymptomatic Hormone Refractory Prostate Cancer
Acronym: KHAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); Dana-Farber Cancer Institute (Other); Sunnybrook Health Sciences Centre (Other); Oregon Health and Science University (Other); M.D. Anderson Cancer Center (Other); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Principal Investigator, Steven Balk, MD, Principle Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-414
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: hormone refractory; KHAD; ketoconazole; dutasteride; hydrocortisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ketoconazole; Hydrocortisone; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KHAD (Experimental): Ketoconazole, Hydrocortisone and Dutasteride Ketoconazole: 200mg orally three times a day on an empty stomach. Hydrocortisone: 30mg in the morning and 10mg in the evening. Dutasteride: 0.5 mg once a day
  Interventions: Drug: Ketoconazole, Hydrocortisone and Dutasteride

INTERVENTIONS:
Drug: Ketoconazole, Hydrocortisone and Dutasteride — Ketoconazole: 200mg orally three times a day on an empty stomach. Hydrocortisone: 30mg in the morning and 10mg in the evening. Pills should be taken with food or milk.
  Dutasteride: 0.5mg orally once a day on an empty stomach or after eating a meal
  Other Names: Dutasteride=Avodart

SUMMARY:
The combination of ketaconazole and hydrocortisone is commonly used for the treatment of prostate cancer. The purpose of this study is to determine if the addition of a drug called dutasteride to this approved combination will make the combination more effective in treating prostate cancer.

DETAILED DESCRIPTION:
* Participants will be seen by the study physician every four weeks and have a short physical examination, blood tests and be asked to provide information about their condition. Every three months they will undergo a bone scan. If the CT scan that was obtained before the participant started the study shows evidence of cancer, they will be asked to repeat this test every three months.
* Ketaconazole will be taken orally three times a day on an empty stomach. Hydrocortisone will be taken orally in the morning and at night. Dutasteride will be taken orally once a day.
* Participants may remain on study drug until there is evidence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented evidence of prostate cancer (needle biopsy or prostatectomy). In the abscence of histologically documented evidence of prostate cancer, the diagnosis must be based on elevated serum PSA and metastatic lesions on bone scan.
* Progressive HRPC defined as a PSA increase over baseline of >25% or 5ng/ml or new lesions on bone/CT scan after conventional androgen deprivation and antiandrogen withdrawal. Evidence of metastatic disease based on positive CT or bone scan is not required.
* PSA of greater than or equal to 2ng/ml and serum total testosterone less than or equal to 50ng/ml
* Prior chemotherapy is permitted if discontinued > 4 weeks prior to starting therapy
* Prior therapy with estrogens is permitted but must have been discontinued > 4 weeks prior to registration
* ECOG Performance Status 0-2
* Adequate renal function, hepatic function, and bone marrow function as outlined in protocol
* ECG showing a normal QT interval

Exclusion Criteria:

* Prior therapy with ketoconazole or corticosteroids for HRPC
* Major surgery or radiation therapy within 4 weeks
* Strontium-89 or samarium-153 therapy within 4 weeks
* Thromboembolism in past 6 months
* Patients who are taking drugs that may further prolong QT intervals and present a known risk for Torsades de Pointes.
* Concomitant use of drugs known to be narrow therapeutic index CTP3A4
* Drugs that are sensitive CYP3A4 substrates
* Alcohol or drug dependence currently or in the last 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-02; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Balk, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (7):
- United States (6):
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oregon Health and Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Sunnybrook and Women's College Health Sciences Center, Toronto, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical oncology clinics
Pre-assignment Details: Required 6 week washout for any AR antagonists
Groups:
- KHAD: KHAD; ketoconazole, hydrocortisone and dutasteride for CRPC
Period: Overall Study
Arm/Group | KHAD
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- KHAD: Ketoconazole, Hydrocortisone and Dutasteride
Arm/Group | KHAD
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 57
Region of Enrollment [Number; unit: participants]
  United States | 49
  Canada | 8

OUTCOME MEASURES:

1. Primary Outcome: PSA Response
Description: PSA decline of 50% from baseline confirmed by a PSA at least 4 weeks later.
Time Frame: From treatment initiation until treatment cessation. Maximum 32 months. Median treament duration 8 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KHAD
Number analyzed (Participants) | 57
percentage of participants | 56 [42.4 to 69.3]

2. Secondary Outcome: Time to Progression
Description: Duration of time from treatment initiation until documented progression (PSA or Disease progression)
Time Frame: Duration of time from treatment initiation until documented progression. Maximum 32 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- KHAD: KHAD: ketoconazole, hydrocortisone and dutasteride for CRPC
Arm/Group | KHAD
Number analyzed (Participants) | 57
months | 14.5 [11 to 17]

ADVERSE EVENTS:
Arm/Group | KHAD
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KHAD (N=57)
grade 4 thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KHAD (N=57)
Hemoglobin (Blood and lymphatic system disorders) | 23
Hematologic-other (Blood and lymphatic system disorders) | 1
Cardiomyopathy, restrictive (Cardiac disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Endocrine-other (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Dry eye syndrome (Eye disorders) | 3
Vision-blurred (Eye disorders) | 2
Tearing (Eye disorders) | 1
Ocular-other (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 4
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 6
Incontinence, anal (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 4
GI-other (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 21
Fever w/o neutropenia (General disorders) | 1
Constitutional, other (General disorders) | 6
Edema head and neck (General disorders) | 1
Edema limb (General disorders) | 10
Pain-other (General disorders) | 5
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Lymphopenia (Investigations) | 3
Weight gain (Investigations) | 2
Alkaline phosphatase (Investigations) | 6
ALT, SGPT (Investigations) | 27
AST, SGOT (Investigations) | 29
Bilirubin (Investigations) | 3
Creatinine (Investigations) | 15
Metabolic/Laboratory-other (Investigations) | 2
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 21
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 6
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Neurologic-other (Nervous system disorders) | 3
Head/headache (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 5
Agitation (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Personality (Psychiatric disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 2
Gynecomastia (Reproductive system and breast disorders) | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 12
Hypotension (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No